CLINICAL TRIAL: NCT05277025
Title: Pain Processing in Inflammatory and Non-Inflammatory Chronic Pain Syndromes
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202200105
Record Dates: First submitted 2022-02-28; First posted 2022-03-14 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia; Rheumatoid Arthritis
MeSH Terms: conditions — Fibromyalgia; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fibromyalgia: Participants who fulfill the 1990 and 2011 American College of Rheumatology Criteria for FM.
- Rheumatoid Arthritis: Participants who fulfill the 2010 American College of Rheumatology (ACR)-European League against rheumatism (EULAR) classification criteria for RA.
- Healthy Volunteers: Participants who do not have significant pain/fatigue/anxiety/depression.

SUMMARY:
Fibromyalgia (FM) is a chronic musculoskeletal pain disorder that afflicts up to 4% of the general population. The evaluation of pain mechanisms in FM has shown predominant central abnormalities and therefore has been designated as nociplastic pain syndrome. Rheumatoid arthritis (RA) is characterized by polyarthritis and pain from inflamed tissues, consistent with nociceptive pain. FM and RA patients may utilize overlapping pain mechanisms resulting in nociceptive and nociplastic pain.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Fulfills the 1990 and 2011 American College of Rheumatology Criteria for FM
* Fulfills the 2010 ACR-EULAR classification criteria for RA
* Healthy volunteers: No significant pain/fatigue/depression/anxiety.

Exclusion Criteria:

* Diabetes
* Cancer
* Advanced liver, kidney or cardiovascular disease
* Neuropathic pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a case-control study of FM, RA and healthy controls (HC) that will be enrolled in a ratio of 1:1:1. Healthy controls will be aged/gender matched to the FM and RA groups.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Thresholds | One hour
  Using an algometer pressure pain thresholds will be obtained several times at the upper and lower extremities

CONTACTS AND LOCATIONS:
Overall Officials: Roland Staud, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States